CLINICAL TRIAL: NCT04745819
Title: Epidemiological Screening of Psychiatric Disorders Among School Aged Children and Adolescent in Assiut Governorate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer, resarcher OF Neurology and Psychiatry department, Assiut University
Other Study IDs: epidemyology study in Assiut
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Child Behavior Disorders; Child Mental Disorder; Adolescent Behaviour
Keywords: child; adolescent; psychiatry
MeSH Terms: conditions — Child Behavior Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: 1. The Child Behavior Checklist (CBCL), parent form — It consists of 113 items; the parents complete it to detect emotional and behavioural problems in children and adolescents aged 6 to 18 years. It is scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). The time duration for item responses is the past six months.

SUMMARY:
Paediatric behavioural, developmental, and mental health issues are more common than childhood cancers, cardiac problems, and renal problems combined.

Behavioural problems have often been conceptualized along two broad spectrums: internalizing problems which are expressed in intrapersonal manifestation, such as anxiety, depression, and withdrawal; and externalizing problems which are demonstrated in interpersonal manifestation, such as hyperactivity and aggression The lack of attention to the mental health of children and adolescents may lead to mental disorders with lifelong consequences, undermines compliance with health regimens, and reduces the capacity of societies to be safe and productive. As, children and adolescent mental health problems often have serious long term debilitating effects . Early identification and treatment of these problems are in the best interest of children, adolescents, their families, and society as a whole . All three essential ways in which epidemiology can contribute to our understanding of children and adolescent mental health: community burden, measurement, and triage were of utmost importance. planning and conducting the survey.

In this study the researchers will present the first large-scale survey of child and adolescent psychiatric disorders at Assiut government For adequate planning of services, including evidence-based mental health prevention and intervention, a population-representative survey of children and adolescent estimating mental disorders was urgently needed

ELIGIBILITY:
Inclusion Criteria:

1. age of children (6-18 years)
2. both males and females.
3. have education in school at Assiut government.

Exclusion Criteria:

1- unwilling parent to recruited in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This is study will take part in the first screening phase in the Assiut government school community study. The other part will be in the child and adolescent psychiatry clinic at Neurology and Psychiatry department at Assiut university hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
measure the prevalence of DSM 5 psychiatric disorders in the community sample of school children in Assiut government. | through study completion, an average of 1 year
measure of risk factor of DSM 5 psychiatric disorders in the community sample of school children in Assiut government. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No